CLINICAL TRIAL: NCT06711055
Title: A Cohort Study of Adjuvant Therapy With Taxane Combined Targeted Therapy for Low-risk HER2 Positive and Lymph Node Negative Breast Cancer
Brief Title: Taxane Combined Targeted Therapy for Low-risk HER2 Positive and Lymph Node Negative Breast Cancer
Acronym: TaxHER
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z164
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: Taxane; target therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Taxanes combined with trastuzumab: Taxane with trastuzumab. Taxane drugs allow the selection of paclitaxel, liposomal paclitaxel, albumin paclitaxel, or docetaxel. Chemotherapy is administered in a single week regimen with 12 cycles or a 3-week regimen with 4 cycles, with target therapy for 1 year

SUMMARY:
Human epidermal growth factor receptor 2 (HER2) positive breast cancer is a molecular subtype with high malignancy and high risk of recurrence and metastasis. HER2 targeted drugs has greatly improved the prognosis and survival of such patients. At present, for HER2 positive breast cancer patients with negative lymph nodes, chemotherapy drugs combined with trastuzumab is the current standard treatment scheme, and in most cases, chemotherapy uses a combination of two drugs, while the main beneficiaries of the trastuzumab and paltuzumab are concentrated in the group of patients with positive lymph nodes. Can targeted therapy be used to reduce the progression of chemotherapy and further achieve efficient and low toxicity strategies. To explore the efficacy and safety of adjuvant therapy of taxane chemotherapy combined with trastuzumab targeting therapy for low-risk HER2 positive and lymph node negative early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) Treatment in Peking University People's Hospital for radical resection of breast cancer and had hospitalization records;
* 2) Postoperative pathology confirmed invasive breast cancer, and the pathological stage was T1a-b (T ≤ 1cm), N0, HER2 positive, with high-risk factors (G3, or hormone receptor negative); Or the pathological stage is T1c (1cm < T ≤ 2cm), N0, and there are no high-risk factors (G1/G2, hormone receptor positive);
* 3)Signed an agreement to participate in the PKUPH Breast Disease Cohort study at Peking University People's Hospital.

Exclusion Criteria:

* 1) Lack of clinical pathological data (such as imaging data, pathological data);
* 2) Preoperative neoadjuvant therapy;
* 3) Patients with metastatic breast cancer or bilateral breast cancer;
* 4) Failed to undergo curative surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: invasive breast cancer, and the pathological stage was T1a-b (T ≤ 1cm), N0, HER2 positive, with high-risk factors (G3, or hormone receptor negative); T1c (1cm < T ≤ 2cm), N0, and there are no high-risk factors (G1/G2, hormone receptor positive)
Sampling Method: Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
invasive disease free survival | 5 years
  The time from enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.

SECONDARY OUTCOMES:
disease free survival | 5 years
  The time from enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.
distant disease free survival | 5 years
  The time from enrollment in the study to the occurrence of distant recurrence and metastasis.
breast cancer specific survival | 5 years
  Time from enrollment to death due to breast cancer. Time from enrollment to death due to breast cancer.
overall survival | 5 years
  The time from enrollment in the study to death caused by any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China